CLINICAL TRIAL: NCT05655065
Title: Effects of Increasing Mean Arterial Pressure on Renal Function in Patients with Shock and with Elevated Central Venous Pressure : a Pilot Study for the Individualization of Mean Arterial Pressure
Brief Title: Effects of Increasing Mean Arterial Pressure on Renal Function in Patients with Shock and with Elevated Central Venous Pressure
Acronym: MAPAKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 49RC22_0293
Record Dates: First submitted 2022-11-03; First posted 2022-12-16 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Shock
Keywords: mean arterial pressure; central venous pressure; Renal function
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Increase of MAP at low target 65-70 mmHg (with catecholamines or volemic expansion) (Active Comparator): Target of mean arterial pressure (MAP) at 65-70 mmHg The therapeutic means used to obtain the MAP objectives within each group (increase in catecholamines and / or volume expansion) are left to the discretion of the clinician, in accordance with the recommendations.
  Interventions: Procedure: increase of mean arterial pressure at 65-70 mmHg
- Increase of MAP at high target 80-85 mmHg (with catecholamines or volemic expansion) (Experimental): Target of mean arterial pressure (MAP) at 80-85 mmHg The therapeutic means used to obtain the MAP objectives within each group (increase in catecholamines and / or volume expansion) are left to the discretion of the clinician, in accordance with the recommendations.
  Interventions: Procedure: increase of mean arterial pressure at 80-85 mmHg

INTERVENTIONS:
Procedure: increase of mean arterial pressure at 65-70 mmHg — Increase of mean arterial pressure at 65-70 mmHg (with catecholamines or volemic expansion at the discretion of the clinician)
  Arms: Increase of MAP at low target 65-70 mmHg (with catecholamines or volemic expansion)
Procedure: increase of mean arterial pressure at 80-85 mmHg — Increase of mean arterial pressure at 80-85mmHg (with catecholamines or volemic expansion at the discretion of the clinician).
  Arms: Increase of MAP at high target 80-85 mmHg (with catecholamines or volemic expansion)

SUMMARY:
The purpose of this study is to assess the effect of a higher mean arterial pressure on renal function for patients with shock and elevated central venous pressure.

DETAILED DESCRIPTION:
Current recommandation for mean arterial pressure (MAP) target is 65 mmHg for septic shock, but optimal target to prevent acute renal failure (ARF) remains unknown.

High central venous pressure (CVP) can lead to acute renal failure through venous congestion , and is associated with acute renal failure in intensive care unit.

A decrease of renal perfusion pressure, defined by MAP - CVP, has been shown to be associated with risk of acute renal failure.

The main objective of this trial is to evaluate if an optimisation of renal perfusion pressure, by a higher MAP when CVP is high (≥ 12 cmH2O), can improve renal function.

In this interventional monocenter trial, each patient will be evaluated during 2 consecutive periods of 6 hours, with a temporary MAP target

* Target at 65-70mmHg during 6 hours
* Target at 80-85mmHg during 6 hours

Patients will be randomized into two groups to define the order of targets. There will be a stratification on previous arterial hypertension. Renal function will be measured at the end of each period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old )
* Arterial hypotension requiring the etablishment of catecholamines
* Norepinephrine dose ⩾ 0.1µg/kg/min at the inclusion
* High central venous pressure ≥ 12mmHg
* Cardiac output monitoring (PICCO or Swan Ganz)

Exclusion Criteria:

* Anuria
* Patient with an emergency indication of renal replacement therapy (severe hyperkalemia, severe metabolical acidosis with pH <7.15, acute pulmonary edema due to fluid overload resulting in severe hypoxemia, serum urea concentration > 40 mmol/l)
* Pregnant, lactating or parturient woman
* Patient deprived of liberty by judicial or administrative decision
* Patient with psychiatric compulsory care
* Patient subject to legal protection measures
* Patients with do-no-reanimate order or withdrawal of life sustaining support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of creatinine clearance | At 6 hours and at 12 hours
  Creatinine clearance is calculated with the formula UV/P as follow :
  * U being the urinary creatinine concentration in μmol/l
  * V the urinary volume expressed in ml per unit time
  * P the plasmatic creatinine concentration in μmol/l

SECONDARY OUTCOMES:
Changes of renal resistive index | At 6 hours and 12 hours
  We will assess the changes of the renal resistive index with a low MAP target (65-70mmHg) and with a high MAP target (80-85mmHg).
  Renal resistive index is measured with the use of doppler sonography and is calculated as follow :
  (peak systolic velocity - end diastolic velocity / peak systolic velocity) Renal resistive index from 3 waveforms are averaged to arrive at mean RI values for each kidney.
Co-morbidities | At inclusion.
  We will report rate of pre-existing conditions : ischemic heart disease, chronic heart failure, chronic obstructive pulmonary disease, chronic kidney disease, chronic kidney disease requiring long-term dialysis, liver cirrhosis, diabetes, cancer or autoimmune disease, chronic arterial hypertension.
Arterial hypertension treatment | At inclusion.
  We will report the anterior use of arterial hypertension treatment.
Introduction time of norepinephrine | At inclusion
  Day and hour of norepinephrine introduction.
Norepinephrine dose | At inclusion, then every hours up to hour 12
  Norepinephrine dose will be recorded every 2 hours during the two periods
Amount of fluids (unit = L ) | At 6 hours and 12 hours
  Amount of fluids received will be recorded at the end of each period.
Quantity of nephrotoxic drugs | At inclusion, at 6 hours and 12 hours
  The quantity of nephrotoxic drugs administrated will be recorded.
Intra-vesical pression | At inclusion then every hour up to 12 hours.
  We will measure intra-vesical pression with the use of urinary catheter.
Number of day with supportive care in intensive care unit (cathecolamines, renal replacement therapy, mechanical ventilation, extracorporeal membrane oxygenation) | Day 90
  Quantification of the number of days with supportive care (catecholamine,renal replacement therapy, mechanical ventilation, extracorporeal membrane oxygenation)
Number of days in intensive care unit | Day 90
  Quantification of the number of days hospitalized in intensive care unit
Number of days in hospital | Day 90
  Quantification of the number of days hospitalized
Survival at day 90 | Day 90
  Status alive or dead at day 90.
Echocardiographic evaluation of left ventricular function | At inclusion, at 6 hours et at 12 hours
  We will report visual estimation of left ventricular ejection fraction (in percent).
Tricuspid annular plane systolic excursion (TAPSE) | At inclusion, at 6 hours and at 12 hours.
  We will report the tricuspid annular plane systolic excursion (mm) measured on echocardiographic to evaluate the right ventricular function.
Right S' wave | At inclusion, at 6 hours and at 12 hours.
  We will report the right S' wave (cm/s) measured on echocardiographic to evaluate the right ventricular function.
Tidal volume | At inclusion, at 6 Horus and at 12 jours
  We will report the tidal volume set on the ventilator.
Plateau pressure | At inclusion, at 6 hours and at 12 Hours.
  We will report the plateau pressure (mmHg) measured on the ventilator.
End-expiratory pressure | At inclusion, at 6 hours and at 12 Hours.
  We will report the end expiratory pressure (mmHg) measured on the ventilator.
Pulmonary compliance | At inclusion, at 6 hours and at 12 Hours.
  The pulmonary compliance (in ml/mmHg) will be calculated using the formula : Pulmonary compliance = Tidal volume / (plateau pressure - end-expiratory pressure).
Cardiac index measured | At inclusion and every hour up to 12 hours.
  We will record the cardiac index measured if the patient is monitored with a Swan Ganz catheter.
Continuous cardiac output | At inclusion and every hour up to 12 hours
  We will record continuous cardiac output monitoring on pulse contour analysis of the invasive arterial blood pressure curve if the patient is monitored with Pulse index Continuous Cardiac Output (PICCO).
Pulmonary pressions | At inclusion and every hour up to 12 hours
  We will record the pulmonary arterial pressions if the patient is monitored with Swan Gan catheter.
Extra vascular lung water | At inclusion and every hour up to 12 hours
  We will record extra vascular lung water if the patient is monitored with PICCO.
Pulmonary Vascular Permeability Indice | At inclusion and every hour up to 12 hours
  We will record Pulmonary Vascular Permeability Indice if the patient is monitored with PICCO.
Troponin | At inclusion, at 6 hours and at 12 hours.
  Troponine dosage at the inclusion and the end of each period.
Collection of all adverse event | At 6 hours and at 12 hours.
  We will collect all adverse event during the protocol.
Ionogram | At inclusion, at 6 hours and at 12 hours.
  Results of ionogram will be recorded.
paO2 | At inclusion, at 6 hours and at 12 hours.
  paO2 measured on blood gases will be recorded (in mmHg).
paCO2 | At inclusion, at 6 hours and at 12 hours.
  paCO2 measured on blood gases will be recorded (in mmHg).
Lactates | At inclusion, at 6 hours and at 12 hours.
  Lactates measured on blood gases will be recorded (in mmol/l).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ASFAR, MD PhD, Principal Investigator — Angers University Hospital
Locations (2):
- France (2):
  - Angers University Hospital, Angers
  - Vendée Hospital, La Roche-sur-Yon